CLINICAL TRIAL: NCT03743818
Title: COMPARATIVE STUDY OF THE EFFICACY OF HYALURONIC ACID, DRY NEEDLING AND COMBINED TREATMENT IN PATELLAR OSTEOARTHRITIS: NON-CONTROLLED RANDOMIZED CLINICAL TRIAL WITH BLINDED EVALUATOR
Brief Title: COMPARATIVE STUDY OF THE EFFICACY OF HYALURONIC ACID, DRY NEEDLING AND COMBINED TREATMENT IN PATELLAR OSTEOARTHRITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Collaborators: Verónica Prieto Domínguez (Unknown); Raúl Vittori (Unknown); Ignacio Normand Farias (Unknown)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCAvila
Record Dates: First submitted 2018-11-11; First posted 2018-11-16 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Dry Needling; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dry needling (Experimental): dry needling in trigger point in vastus medialis of quadriceps
  Interventions: Device: dry needling
- standardized treatment protocol (Active Comparator): in the standardized treatment protocol the investigators including ultrasound, tens, and isometric quadriceps contractions
  Interventions: Other: ultrasound
- hialuronic acid (Active Comparator): infiltration of hyaluronic acid in the affected knee
  Interventions: Device: hyauluronic acid

INTERVENTIONS:
Device: dry needling — dry needling on the trigger point of the vastus medialis of the quadriceps
  Arms: dry needling
Other: ultrasound — aply ultrasound on the knee
  Arms: standardized treatment protocol
Device: hyauluronic acid — aply hyaluronic acid on the knee
  Arms: hialuronic acid

SUMMARY:
Randomized clinical trial in patients with knee osteoarthritis. Sixty patients will be evaluated, divided in three groups (20 in each). One group A will be treated by dry needling in the vast internal, other group B will be treated with a standardized treatment protocol (electrotherapy and manual therapy), and group C will be treated with hialuronic acid. The investigators want to observe which technique is the most effective in osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee pain and diagnosed of osteoarthritis knee and confirm RNM
* More 18 years.
* Less 55 years

Exclusion Criteria:

* More 55 years.
* Less 18 years.
* mental dysfunction
* those who have any type of complication that can cause myofascial or neuropathic pain in the lower limb, such as lumbo-sacral radiculopathy, neuropraxia, neurothymesis, axonotmesis, or meralgia paraesthetica; who have any condition generally considered to be a factor in perpetuating TrPs, such as fibromyalgia, hypothyroidism, or iron deficiency; and patients who may have a fear of needles (belonephobia) will be excluded.

Patients with lower limb dysmetries of 0.50 cm or more were also excluded from this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 month
  Pain 0 maximum pain score---------10 minimum pain score

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC scale) | 1 month
  scale with questions to mesure pain,(5 questions), stiffness (2 questions) and physical function (17 questions). There are five answers in each questions: none, mild, moderate, severe and extreme.
International Physical Activity Questionnaire scale | 1 month
  questions to mesure physical activity. 7 questions about the time that employed the patients in activities physical ( hours/day, minutes/day, days/week or any activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Fisiosalud Avila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Velazquez-Saornil J, Ruiz-Ruiz B, Rodriguez-Sanz D, Romero-Morales C, Lopez-Lopez D, Calvo-Lobo C. Efficacy of quadriceps vastus medialis dry needling in a rehabilitation protocol after surgical reconstruction of complete anterior cruciate ligament rupture. Medicine (Baltimore). 2017 Apr;96(17):e6726. doi: 10.1097/MD.0000000000006726. PMID 28445290
- [Result] Sanchez-Romero EA, Pecos-Martin D, Calvo-Lobo C, Ochoa-Saez V, Burgos-Caballero V, Fernandez-Carnero J. Effects of dry needling in an exercise program for older adults with knee osteoarthritis: A pilot clinical trial. Medicine (Baltimore). 2018 Jun;97(26):e11255. doi: 10.1097/MD.0000000000011255. PMID 29952993
- [Result] Espi-Lopez GV, Serra-Ano P, Vicent-Ferrando J, Sanchez-Moreno-Giner M, Arias-Buria JL, Cleland J, Fernandez-de-Las-Penas C. Effectiveness of Inclusion of Dry Needling in a Multimodal Therapy Program for Patellofemoral Pain: A Randomized Parallel-Group Trial. J Orthop Sports Phys Ther. 2017 Jun;47(6):392-401. doi: 10.2519/jospt.2017.7389. Epub 2017 May 13. PMID 28504067
- [Result] Mayoral O, Salvat I, Martin MT, Martin S, Santiago J, Cotarelo J, Rodriguez C. Efficacy of myofascial trigger point dry needling in the prevention of pain after total knee arthroplasty: a randomized, double-blinded, placebo-controlled trial. Evid Based Complement Alternat Med. 2013;2013:694941. doi: 10.1155/2013/694941. Epub 2013 Mar 27. PMID 23606888